CLINICAL TRIAL: NCT00994136
Title: Locking of Totally Implanted Venous Access Devices and Tunneled Catheters With or Without Heparin: a Randomised Open-labeled Controlled Trial
Brief Title: Safety of Catheter Lock With or Without Heparin in Implanted Central Venous Catheters
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Leuvens Kanker Instituut (Unknown)
Responsible Party: Marguerite Stas, Universitaire Ziekenhuizen Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SM008
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-06

CONDITIONS: Oncology, Medical; Hematologic Disease
Keywords: Catheters, indwelling; Catheterization, Central Venous; Withdrawal occlusion; Heparin lock
MeSH Terms: conditions — Neoplasms; Hematologic Diseases | interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal saline (Experimental): In the intervention group the use of heparin as locking solution in the catheter lumen (or lumina) when the catheter is not longer in use is omitted. Catheters are locked under positive pressure with normal saline in stead injecting an extra volume of heparinised saline (100IU/ml).
  Interventions: Drug: normal saline
- Heparin lock (No Intervention)
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: normal saline — Ten milliliters of normal saline will be injected at the end of the intravenous therapy. Injection is performed with the start/stop method and with the positive pressure technique (clamping the catheter while injecting the last milliliters of normal saline)

SUMMARY:
Long-term central venous access devices are considered as safe for the administration of medication as chemotherapy, but are also used for blood sampling. For years these catheters have been locked with a heparin solution in order to avoid occlusion. However, no scientific evidence supports heparin locking when the device is not in use. Advanced technology as needleless caps and valved catheters and port reservoirs confirms this trend to use 'saline only' for locking these devices. Therefore the investigators hypothesize is that there will be no difference in proportion of occlusions and catheter related bacteremia in long-term venous access devices locked with 'saline only' versus with heparin.

ELIGIBILITY:
Inclusion Criteria:

* Oncology and hematology patients
* Life expectancy of minimum of 180 days

Exclusion Criteria:

* second or femoral long-term central venous access device
* known allergy to heparin (HIT)
* coagulation disorders(INR >2, Blood platelets > 1,000,000/mm3)
* therapeutic intravenous heparin administration

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Withdrawal occlusion | within180 days

SECONDARY OUTCOMES:
all catheter-related bacteremia | within 180 days
Incidence of functional problems other than withdrawal occlusion | within 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Marguerite Stas, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Universitaire Ziekenhuizen Leuven, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Background] Stephens LC, Haire WD, Tarantolo S, Reed E, Schmit-Pokorny K, Kessinger A, Klein R. Normal saline versus heparin flush for maintaining central venous catheter patency during apheresis collection of peripheral blood stem cells (PBSC). Transfus Sci. 1997 Jun;18(2):187-93. doi: 10.1016/s0955-3886(97)00008-8. PMID 10174683
- [Background] Kadidal VV, Mayo DJ, Horne MK. Heparin-induced thrombocytopenia (HIT) due to heparin flushes: a report of three cases. J Intern Med. 1999 Sep;246(3):325-9. doi: 10.1046/j.1365-2796.1999.00527.x. PMID 10476001
- [Background] Rama BN, Haake RE, Bander SJ, Ghasem-Zadeh A, Gorla C. Heparin-flush associated thrombocytopenia--induced hemorrhage: a case report. Nebr Med J. 1991 Dec;76(12):392-4. PMID 1784321
- [Background] Bazelly B, Lotz JP, Milleron B. [The maintenance of totally implantable perfusion sites]. Rev Pneumol Clin. 1994;50(1):43-4. No abstract available. French. PMID 7973333
- [Background] Randolph AG, Cook DJ, Gonzales CA, Andrew M. Benefit of heparin in peripheral venous and arterial catheters: systematic review and meta-analysis of randomised controlled trials. BMJ. 1998 Mar 28;316(7136):969-75. doi: 10.1136/bmj.316.7136.969. PMID 9550955
- [Background] Theard JL, Robard S. [Outcome of usage protocols on implantable devices]. Ann Fr Anesth Reanim. 1995;14(6):534-5. doi: 10.1016/s0750-7658(05)80501-5. No abstract available. French. PMID 8745984
- [Background] Smith S, Dawson S, Hennessey R, Andrew M. Maintenance of the patency of indwelling central venous catheters: is heparin necessary? Am J Pediatr Hematol Oncol. 1991 Summer;13(2):141-3. doi: 10.1097/00043426-199122000-00005. PMID 2069221
- [Background] Brown-Smith JK, Stoner MH, Barley ZA. Tunneled catheter thrombosis: factors related to incidence. Oncol Nurs Forum. 1990 Jul-Aug;17(4):543-9. PMID 2399167
- [Background] Kelly C, Dumenko L, McGregor SE, McHutchion ME. A change in flushing protocols of central venous catheters. Oncol Nurs Forum. 1992 May;19(4):599-605. PMID 1603675
- [Background] Goossens GA, Verbeeck G, Moons P, Sermeus W, De Wever I, Stas M. Functional evaluation of conventional 'Celsite' venous ports versus 'Vortex' ports with a tangential outlet: a prospective randomised pilot study. Support Care Cancer. 2008 Dec;16(12):1367-74. doi: 10.1007/s00520-008-0436-y. Epub 2008 Apr 15. PMID 18414904
- [Background] McDiarmid S, Hamelin L, Huebsch LB. Leading change: Retrospective evaluation of a nurse-led initiative in vascular access options for autologous stem cell transplant recipients ranging from Hickman catheters to peripherally inserted central catheters. J Infus Nurs. 2006 Mar-Apr;29(2):81-8. doi: 10.1097/00129804-200603000-00005. PMID 16569997
- [Background] Horan TC, Andrus M, Dudeck MA. CDC/NHSN surveillance definition of health care-associated infection and criteria for specific types of infections in the acute care setting. Am J Infect Control. 2008 Jun;36(5):309-32. doi: 10.1016/j.ajic.2008.03.002. No abstract available. PMID 18538699
- [Background] Caers J, Fontaine C, Vinh-Hung V, De Mey J, Ponnet G, Oost C, Lamote J, De Greve J, Van Camp B, Lacor P. Catheter tip position as a risk factor for thrombosis associated with the use of subcutaneous infusion ports. Support Care Cancer. 2005 May;13(5):325-31. doi: 10.1007/s00520-004-0723-1. Epub 2004 Nov 5. PMID 15538639
- [Background] Petersen J, Delaney JH, Brakstad MT, Rowbotham RK, Bagley CM Jr. Silicone venous access devices positioned with their tips high in the superior vena cava are more likely to malfunction. Am J Surg. 1999 Jul;178(1):38-41. doi: 10.1016/s0002-9610(99)00124-5. PMID 10456700
- [Background] Brouns F, Schuermans A, Verhaegen J, De Wever I, Stas M. Infection assessment of totally implanted long-term venous access devices. J Vasc Access. 2006 Jan-Mar;7(1):24-8. doi: 10.1177/112972980600700105. PMID 16596525
- [Background] Hadaway LC. Flushing to reduce central catheter occlusions. Nursing. 2000 Oct;30(10):74. doi: 10.1097/00152193-200030100-00037. No abstract available. PMID 11096978
- [Background] Ryder M. The role of biofilm in vascular catheter-related infections. 15-25. 2001. Ref Type: Serial (Book,Monograph)
- [Background] Cossey V, Thelissen MJ, Goossens GA, Stas M, Schuermans A. Needleless positive-pressure mechanical valve connectors: are they safe? Clin Microbiol Infect 2008;S121-666.doi:10.1111/j.1469-0691.2008.02007.x.